CLINICAL TRIAL: NCT00833781
Title: A Pilot, Double-blind, Placebo-controlled, Randomized Clinical Trial of mRNA-transfected Autologous Dendritic Cells in Subjects With Well-controlled Chronic HIV-1 Infection on Highly Active Antiretroviral Therapy
Brief Title: A Pilot Study of a Dendritic Cell Vaccine in HIV-1 Infected Subjects
Acronym: PARC002
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Rajesh T. Gandhi, MD, Director of Education, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008p001577; R01AI066992-04 (NIH); DAIDS-ES ID 10731 (Other: DAIDS)
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: HIV-1 Infection; HIV Infections
Keywords: HIV vaccine; Dendritic cells; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — RNA, Messenger

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mRNA-transfected dendritic cells (Active Comparator): Participants in this arm/group received mRNA-transfected autologous dendritic cells
  Interventions: Biological: mRNA-transfected autologous dendritic cells
- Dendritic cells without mRNA (Placebo Comparator): Participants in this arm/group received autologous dendritic cells with no mRNA transfection
  Interventions: Biological: autologous dendritic cells with no mRNA transfection

INTERVENTIONS:
Biological: mRNA-transfected autologous dendritic cells — Injections will be administered intradermally at weeks 0, 2, 6 and 10.
  Arms: mRNA-transfected dendritic cells
Biological: autologous dendritic cells with no mRNA transfection — Injections will be administered intradermally at weeks 0, 2, 6 and 10.
  Other Names: Autologous dendritic cells not transfected with mRNA.
  Arms: Dendritic cells without mRNA

SUMMARY:
The purpose of the study is to find out whether an experimental autologous dendritic cell vaccine is safe, well tolerated, and whether it can strengthen the immune system's response to HIV.

DETAILED DESCRIPTION:
This is a randomized trial to evaluate whether mRNA-transfected dendritic cell vaccination is safe and immunogenic in HIV-infected participants who are on antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive
* CD4+ T Cell count >200
* Undetectable HIV viral load for 6 months prior to screening
* On antiretroviral treatment for 12 months prior to screening

Exclusion Criteria:

* Hepatitis C positive
* Detectable HIV viral load within 6 months prior to study entry
* Females who are pregnant or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Gandhi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Infectious Disease Unit; Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gandhi RT, Kwon DS, Macklin EA, Shopis JR, McLean AP, McBrine N, Flynn T, Peter L, Sbrolla A, Kaufmann DE, Porichis F, Walker BD, Bhardwaj N, Barouch DH, Kavanagh DG. Immunization of HIV-1-Infected Persons With Autologous Dendritic Cells Transfected With mRNA Encoding HIV-1 Gag and Nef: Results of a Randomized, Placebo-Controlled Clinical Trial. J Acquir Immune Defic Syndr. 2016 Mar 1;71(3):246-53. doi: 10.1097/QAI.0000000000000852. PMID 26379068

RESULTS

PARTICIPANT FLOW:
Groups:
- mRNA-transfected Autologous Dendritic Cell Vaccine.: mRNA-transfected autologous dendritic cells: Injections will be administered intradermally at weeks 0, 2, 6 and 10.
- Autologous Dendritic Cells Without Transfected mRNA.: Dendritic cell vaccine without transfected mRNA.
  Autologous dendritic cells not transfected with mRNA.: Injections will be administered intradermally at weeks 0, 2, 6 and 10.
Period: Overall Study
Arm/Group | mRNA-transfected Autologous Dendritic Cell Vaccine. | Autologous Dendritic Cells Without Transfected mRNA.
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mRNA-transfected Autologous Dendritic Cell Vaccine. | Autologous Dendritic Cells Without Transfected mRNA. | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Median (Full Range); unit: years] | 44 [33 to 55] | 49 [42 to 52] | 46.7 [33 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Safety of the DC Vaccine (as Measured by Frequency of Adverse Events)
Description: Number of participants with grade 3 or 4 adverse events related to vaccination
Time Frame: After vaccination
Measure: Number; unit: participants
Groups:
- mRNA-transfected Autologous Dendritic Cells; Dendritic Cell Vaccine Without Transfected mRNA.: Injections were administered intradermally at weeks 0, 2, 6 and 10.
Arm/Group | mRNA-transfected Autologous Dendritic Cells | Dendritic Cell Vaccine Without Transfected mRNA.
Number analyzed (Participants) | 10 | 5
participants | 0 | 0

2. Secondary Outcome: T Cell Proliferation
Time Frame: Baseline to week 14
Measure: Mean (95% Confidence Interval); unit: fold change
Arm/Group | mRNA-transfected Autologous Dendritic Cells | Dendritic Cell Vaccine Without Transfected mRNA.
Number analyzed (Participants) | 10 | 5
fold change
  CD4 Gag proliferative response | 2.465 [1.167 to 5.208] | 0.717 [0.253 to 2.033]
  CD4 Nef Proliferative response | 2.292 [1.044 to 5.035] | 0.363 [0.12 to 1.102]

3. Primary Outcome: Change From Baseline to Week 14 in ELISPOT Response to Gag and Nef
Description: Immunogenicity was measure by interferon gamma enzyme-linked immunospot (ELISPOT) assay. The number of spot forming cells per million PBMC was determined at each time point. The fold ratio represents week 14 value divided by value at baseline.
Time Frame: Baseline and 14 weeks
Measure: Median (Full Range); unit: fold ratio
Arm/Group | mRNA-transfected Autologous Dendritic Cells | Dendritic Cell Vaccine Without Transfected mRNA.
Number analyzed (Participants) | 10 | 5
fold ratio
  Gag ELISPOT | 1.06 [0.893 to 1.259] | 1.058 [0.836 to 1.33]
  Nef ELISPOT | 1.15 [0.979 to 1.351] | 1.021 [0.813 to 1.281]

4. Secondary Outcome: IL2 and IFN Gamma Production
Time Frame: Baseline to week 14
Population: Results from these assays were too variable to be interpretable.
Arm/Group | mRNA-transfected Autologous Dendritic Cells | Dendritic Cell Vaccine Without Transfected mRNA.
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | mRNA Transfected DCs
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
The trial size is small, precluding detection of small effect sizes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes